CLINICAL TRIAL: NCT05192265
Title: Comparative Efficacy and Safety of Pyronaridine-Artesunate Versus Artemether-Lumefantrine in The Treatment of Acute Uncomplicated Malaria Among Children In South-West Nigeria
Brief Title: Efficacy and Safety of Pyronaridine-Artesunate Versus Artemether-Lumefantrine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Ibadan (Other)
Collaborators: Shin Poong Pharm Co Ltd 161 yoksam-ro, Gangnam-Gu Seoul 135-925, Korea (Unknown); Institute for Advanced Medical Research and Training, University of Ibadan, Ibadan (Unknown)
Responsible Party: Principal Investigator, Adebola E. Orimadegun, Professor, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UI/EC/19/0114
Record Dates: First submitted 2021-12-21; First posted 2022-01-14 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Malaria Fever; Plasmodium Falciparum Malaria; Uncomplicated Malaria
Keywords: Antimalarial; Pyronaridine-artesunate; Artemether-lumefantrine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Antimalarials; pyronaridine tetraphosphate, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Study participants were assigned into one of the two treatment groups according to a pre-generated randomization code. Children randomized to Pyramax™ received three doses of pyronaridine-artesunate granules or tablets manufactured by Shin Poong Pharmaceuticals, Seoul, Korea depending on their body weights. Pyramax granules come in sachets with each containing 60mg of pyronaridine/20mg of artesunate while Pyramax tablets contain 180mg pyronaridine/60mg artesunate. Study participants randomized to Coartem™ received the standard six-dose regimen of AL dispersible tablets (Coartem™, Novartis pharma) twice daily according to body weights.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyramax™ (Experimental): Artesunate-pyronaridine is indicated for the blood-stage treatment of the two dominant strains of malaria: P. falciparum and P. vivax. The medicine is also available in a child-friendly granule formulation to enhance palatability in this vulnerable population. Dosing was administered according to body weight: 5 - <8kg - one sachet daily for 3 days; 8 - <15Kg - two sachets daily for 3 days; 15 - <20 Kg - three sachets daily for 3 days; 20 - <24 Kg - one tablet daily for 3 days; and 24 - <45 Kg - two tablets daily for 3 days.
  Interventions: Drug: Antimalarials, pyronaridine-artesunate
- Coartem™ (Active Comparator): We used the standard six-dose regimen of artemether-lumefantrine dispersible tablets twice daily according to body weights. Each dispersible tablet contains 20mg of artemether/120mg of lumefantrine) and the patients were dosed as follows: 5 -<15Kg one tablet, 15 - <25 Kg two tablets, 25 - <35 Kg three tablets, and ≥35 Kg four tablets at the following dosing intervals:
  * 0 hour - 1st dose;
  * 8 hours - 2nd dose;
  * 24 hours - 3rd dose;
  * 36 hours - 4th dose;
  * 48 hours - 5th dose
  * 60 hours - 6th dose.
  Interventions: Drug: Antimalarials, Artemether + Lumefantrine

INTERVENTIONS:
Drug: Antimalarials, pyronaridine-artesunate — The main interventions investigated are pyronaridine-artesunate granules or tablets (Pyramax™) manufactured by Shin Poong Pharmaceuticals, Seoul, Korea. Pyramax granules come in sachets with each containing 60mg of pyronaridine/20mg of artesunate while Pyramax tablets contain 180mg pyronaridine/60mg artesunate.
  Other Names: Pyramax™
  Arms: Pyramax™
Drug: Antimalarials, Artemether + Lumefantrine — Artemether-lumefantrine dispersible tablets (Coartem™, Novartis pharma) twice daily according to body weights. Each dispersible tablet of AL contains 20mg of artemether/120mg of lumefantrine).
  Other Names: Coartem™, Novartis pharma
  Arms: Coartem™

SUMMARY:
In Nigeria, malaria is the commonest reason for outpatient clinic attendance in childhood and is responsible for about 20% of childhood deaths. The emergence of strains of P. falciparum resistant to chloroquine and sulfadoxine-pyrimethamine led to severe worsening of morbidity and mortality from malaria. As a result of resistance to previously used monotherapy, the World Health Organization (WHO) in 2001, recommended that malaria-endemic countries experiencing drug-resistant malaria infection adopt combination therapy. Artemisinin-based combination therapy (ACT) is preferred to the non-ACT combination. In this randomized open-label clinical trial, the safety and efficacy of pyronaridine-artesunate and artemether-lumefantrine in the treatment of malaria among children aged 3 to 144 months who have microscopically confirmed symptomatic Plasmodium falciparum malaria were compared. The study was carried out at the Oni Memorial Children's Hospital, Ring Road Ibadan. One hundred and seventy-two children between 3 and 120 months who meet the inclusion criteria will be enrolled after obtaining written or witnessed signed informed consent from the parents or guardian. A detailed history and physical examination were carried out on each enrollee. Finger prick blood samples were taken from each enrolee for thick blood smear for malaria parasite, haematocrit, and blood spots on filter paper. Five millilitres of venous blood will be taken from an arm vein for baseline liver function tests, creatinine, and random blood glucose on days 0, 3, 7 and 28. Enrollees were randomized into one of two groups. Group one received pyronaridine-artesunate while group two received artemether-lumefantrine at standard doses. Enrollees were seen daily from days 0-3, and on days 7, 14, 21 and 28. Study drugs were administered supervised at standard dosage on days 0, 1, and 2. History taking, physical examination and blood smears were done at each contact time. Special attention will be paid to adverse effects. Parasite clearance time, fever clearance time and cure rates were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of either gender between the ages of 3months (but weight ≥5 kg) and 12 years who present with symptoms compatible with acute uncomplicated malaria
2. Minimum asexual parasite density of 1000/µl. This will be done at enrolment for all study participants.
3. Fever with an axillary temperature≥ 37.5°C or history of fever within 24hours of presentation
4. Residence within 15 kilometres to the study site.
5. Ability to take drugs orally.
6. Absence of history of ACT intake in the two weeks prior to enrolment
7. A signed informed consent from parents or guardians of the prospective enrollee to participate in the study

Exclusion Criteria:

1. History of allergy to study drugs i.e. artemisinins, lumefantrine and pyronaridine
2. Any concurrent illness that could hamper evaluation of response e.g. bacterial infections, viral infections, severe gastrointestinal disease, malnutrition (weight for height <70%).
3. Presence of clinical evidence of severe malaria such as prostration, inability to drink or breastfeed, persistent vomiting, convulsion, severe anaemia haemoglobin <5 g/dl), unarousable coma
4. Patients with known chronic diseases like chronic kidney disease, chronic liver disease, malnutrition, cardiac failure, Sickle Cell haemoglobin (HbSS) etc.
5. Mixed or mono-infection with another Plasmodium species detected by microscopy;
6. presence of severe malnutrition defined as a child aged between 6-60 months whose weight-for-high is below -3 z-score, or has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 115 mm).
7. Parent or guardian who in the judgment of the investigator will not comply with protocol in the opinion of the investigator

Ages: 3 Months to 144 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
PCR-adjusted adequate clinical and parasitological response (ACPR) | Treatment day 3 to 28
  Defined as absence of patent parasitaemia, regardless of axillary temperature and without evidence of previous treatment failure up to day 28.

SECONDARY OUTCOMES:
Adequate clinical and parasitological response without correction for reinfection | day 28
  Adequate clinical and parasitological response (ACPR; absence of parasitaemia on day 28 without previously meeting criteria for ETF, LCF, or LPF).
  Note:
  ETF: Early treatment failure defined as danger signs or complicated malaria or failure to adequately respond to therapy on days 0-3.
  LCF: Late clinical failure defined as danger signs or complicated malaria or fever and parasitaemia on days 4-28 without previously meeting criteria for ETF or LPF.
  LPF: Late parasitological failure defined as asymptomatic parasitaemia on days 7-28 without previously meeting criteria for ETF or LCF.
Parasite clearance time | Treatment day 0 to 28
  Time from first dose of ACT until first total and continued disappearance of asexual parasite forms.
Fever clearance time | Treatment day 0 to 28
  Time from first dose until the first time the body temperature (for those with a raised temperature at enrolment) decrease to below 37.5 degree Celsius and remain so for at least 24 hours.
Gametocyte carriage | Treatment day 0 to 28
  Proportions of patients with gametocyte at a given point in time.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine O Falade, MB.BS, MSc, FMCP, FWACP, MD, Principal Investigator — University of Ibadan; Consultant Clinical Pharmacologist, University College Hospital, Ibadan
Locations (1):
- Ikeoluwapo O Ajayi, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falade CO, Orimadegun AE, Olusola FI, Michael OS, Anjorin OE, Funwei RI, Adedapo AD, Olusanya AL, Orimadegun BE, Mokuolu OA. Efficacy and safety of pyronaridine-artesunate versus artemether-lumefantrine in the treatment of acute uncomplicated malaria in children in South-West Nigeria: an open-labelled randomized controlled trial. Malar J. 2023 May 13;22(1):154. doi: 10.1186/s12936-023-04574-7. PMID 37179349

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT05192265/Prot_SAP_ICF_001.pdf